CLINICAL TRIAL: NCT00876343
Title: Placebo-Controlled, Double-Blind, Parallel Group-Comparison Study of Aripiprazole as an Adjunctive Therapy in Patients With Major Depressive Disorder
Brief Title: Study of Aripiprazole as an Adjunctive Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-08-001; JapicCTI-090724
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Fixed dose
  Interventions: Drug: Aripiprazole (Fixed dose)
- 2 (Experimental): Titration dose
  Interventions: Drug: Aripiprazole (Titrated dose)
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole (Fixed dose) — administered orally once daily, 3 mg daily, 6 weeks
  Other Names: Aripiprazole
  Arms: 1
Drug: Aripiprazole (Titrated dose) — administered orally once daily, 3 to 15 mg daily, 6 weeks
  Other Names: Aripiprazole
  Arms: 2
Drug: Placebo — administered orally once daily, 6 weeks
  Other Names: Placebo of aripiprazole
  Arms: 3

SUMMARY:
To examine the efficacy and safety of aripiprazole versus placebo as an adjunctive therapy co-administered with either an selective serotonin reuptake inhibitor (SSRI) or a serotonin-norepinephrine reuptake inhibitor (SNRI) in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are either inpatients or outpatients
2. Patients who have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial
3. Patients diagnosed as having either "296.2x Major Depressive Disorder, Single Episode" or "296.3x Major Depressive Disorder, Recurrent" according to DSM-IV-TR, and for whom the current episode of major depressive disorder has been ongoing for more than 8 weeks
4. Patients with a HAM-D17 total score of 18 or more

Exclusion Criteria:

1. Female patients of child bearing potential who wish to become pregnant during the treatment period, or within 4 weeks after study completion/discontinuation
2. Female patients who are pregnant, possibly pregnant, or breast feeding
3. Patients judged to be unable to tolerate any type of antidpressant treatment (including drugs not being used in the current episode of major depressive disorder), based on treatment history to date
4. Patients who have previously received electro-convulsive therapy
5. Patients who have participated in clinical studies on medical devices or other drugs within the past month
6. Patients at risk of having serious adverse events or developing symptoms that could interfere with safety and efficacy evaluations (such as symptoms of fibromyalgia syndrome overlapping with symptoms of depression), based on previous medical history
7. Patients with a history or a complication of diabetes
8. Patients with thyroid disease (excluding patients who are stabilized on drug therapy for at least 3 months)
9. Patients with a history of serotonin syndrome or psychotropic neuroleptic malignant syndrome
10. Patients with a history of seizure disorder (epilepsy etc.)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — OPC-J
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Derived] Ozaki N, Otsubo T, Kato M, Higuchi T, Ono H, Kamijima K; ADMIRE Study Group. Efficacy of aripiprazole augmentation in Japanese patients with major depressive disorder: a subgroup analysis and Montgomery-Asberg Depression Rating Scale and Hamilton Rating Scale for Depression item analyses of the Aripiprazole Depression Multicenter Efficacy study. Psychiatry Clin Neurosci. 2015 Jan;69(1):34-42. doi: 10.1111/pcn.12214. Epub 2014 Aug 4. PMID 24965202
- [Derived] Kamijima K, Higuchi T, Ishigooka J, Ohmori T, Ozaki N, Kanba S, Kinoshita T, Koyama T; ADMIRE Study Group. Aripiprazole augmentation to antidepressant therapy in Japanese patients with major depressive disorder: a randomized, double-blind, placebo-controlled study (ADMIRE study). J Affect Disord. 2013 Dec;151(3):899-905. doi: 10.1016/j.jad.2013.07.035. Epub 2013 Aug 28. PMID 24074484

RESULTS

PARTICIPANT FLOW:
Groups:
- Variable Dose Group of Aripiprazole: Aripiprazole 3~15 mg were administered orally once daily. During the first week, 3 mg was administered once daily. Thereafter, each week, a dose increase of 3 mg per day was carried out
- Fixed Dose Group of Aripiprazole: Aripiprazole 3 mg were administered orally once daily
- Placebo Group: Placebo were administered orally once daily
Period: Overall Study
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group
Started | 194 | 197 | 195
Completed | 177 | 180 | 183
Not Completed | 17 | 17 | 12
Not completed — Adverse Event | 7 | 8 | 2
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 4 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Diabetic glucose level or HbA1C>=6.5% | 0 | 1 | 1
Not completed — Change of residence or other commitments | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group | Total
Number analyzed (Participants) | 194 | 197 | 195 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.6) | 39.2 (9.1) | 38.7 (9.2) | 38.7 (9.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 194 | 197 | 195 | 586
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 73 | 80 | 246
  Male | 101 | 124 | 115 | 340
Region of Enrollment [Number; unit: participants]
  Japan | 194 | 197 | 195 | 586

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The change in MADRS total score from the end of the SSRI/SNRI treatment period to Week 6 of the placebo-controlled, double-blind treatment period by covariance analysis, and compared the aripiprazole variable dose group with the placebo group as well as the aripiprazole fixed dose group with the placebo group.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  The questionnaire includes questions on the following symptoms
  1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
Time Frame: Baseline (the end of the SSRI/SNRI treatment period), at completion of administration
Measure: Mean (Standard Error); unit: Rating score
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group
Number analyzed (Participants) | 194 | 197 | 195
Rating score | -9.6 (0.6) | -10.5 (0.6) | -7.4 (0.6)
Statistical Analysis 1: Comparison: Variable Dose Group of Aripiprazole vs Placebo Group; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.7 to -0.6]
Statistical Analysis 2: Comparison: Fixed Dose Group of Aripiprazole vs Placebo Group; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-4.6 to -1.5]

2. Secondary Outcome: MADRS Response Rate
Description: The percentage of subjects with a decrease in MADRS total score of 50% or more, from the end of the SSRI/SNRI treatment period to the end of the placebo-controlled, double-blind treatment period (or withdrawal).
Time Frame: Baseline (the end of the SSRI/SNRI treatment period), at completion of administration
Measure: Number; unit: percentage of subjects
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group
Number analyzed (Participants) | 194 | 197 | 195
percentage of subjects | 39.2 | 42.1 | 28.2

3. Secondary Outcome: Mean Change in Sheehan Disability Scale (SDISS)
Description: The endpoint evaluated the change in SDISS from the end of the SSRI/SNRI treatment period to Week 6 of the placebo-controlled, double-blind treatment period.
  The patient rates the extent to which his or her 1) work, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline (the end of the SSRI/SNRI treatment period), at completion of administration
Measure: Mean (Standard Error); unit: Rating score
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group
Number analyzed (Participants) | 194 | 197 | 195
Rating score | -1.03 (0.11) | -0.96 (0.11) | -0.46 (0.11)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Variable Dose Group of Aripiprazole | Fixed Dose Group of Aripiprazole | Placebo Group
Serious Adverse Events (participants affected / at risk) | 3/194 | 2/197 | 2/195
Other Adverse Events (participants affected / at risk) | 140/194 | 122/197 | 92/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Variable Dose Group of Aripiprazole (N=194) | Fixed Dose Group of Aripiprazole (N=197) | Placebo Group (N=195)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Variable Dose Group of Aripiprazole (N=194) | Fixed Dose Group of Aripiprazole (N=197) | Placebo Group (N=195)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 15 (15) | 7 (7) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 6 (6) | 10 (10)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (10) | 10 (10)
Salivary Hypersecretion (Gastrointestinal disorders) | 8 (8) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (6) | 3 (3)
Malaise (General disorders) | 10 (10) | 2 (2) | 8 (8)
Oedema Peripheral (General disorders) | 4 (4) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1) | 0 (0)
Thirst (General disorders) | 13 (13) | 10 (10) | 3 (3)
Nasopharyngitis (Infections and infestations) | 31 (32) | 30 (31) | 28 (31)
Alanine Aminotransferase Increased (Investigations) | 13 (13) | 14 (14) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 8 (8) | 10 (10) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 4 (4) | 2 (2) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 6 (6) | 10 (10) | 0 (0)
Blood Pressure Increased (Investigations) | 3 (3) | 5 (5) | 3 (3)
Blood Triglycerides Increased (Investigations) | 8 (9) | 4 (4) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 5 (5) | 6 (6) | 1 (1)
Weight Increased (Investigations) | 12 (12) | 8 (8) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 3 (3)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 4 (4)
Akathisia (Nervous system disorders) | 71 (73) | 28 (30) | 8 (8)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 6 (6)
Dyskinesia (Nervous system disorders) | 2 (2) | 5 (6) | 1 (1)
Dystonia (Nervous system disorders) | 6 (6) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 9 (9) | 15 (16)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Parkinsonism (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 15 (15) | 19 (19) | 13 (14)
Tremor (Nervous system disorders) | 20 (23) | 14 (16) | 5 (5)
Insomnia (Psychiatric disorders) | 10 (10) | 8 (8) | 3 (3)
Terminal Insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No